CLINICAL TRIAL: NCT00732407
Title: Effect of Aliskiren on Arterial Stiffness and Platelet Function in Patients With Type 2 Diabetes Mellitus, a Comparison With Losartan
Brief Title: Aliskiren's Effect on Arterial Stiffness and Platelet Function in Patients With Diabetes Mellitus (DM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Koren Peleg Ronit MD, Assaf-Harofeh Medical Center internal medicine A
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: ronit2
Record Dates: First submitted 2008-08-10; First posted 2008-08-12 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Diabetes Mellitus; Atherosclerosis
Keywords: aliskiren; arteial stiffness; platelet function; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Atherosclerosis | interventions — aliskiren; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients with diabetes melittus treated with an ACE inhibitor will be treated with aliskiren
  Interventions: Drug: aliskiren; Drug: losartan
- 2 (Experimental): Patients with diabetes melittus treated with an ACE inhibitor will be given losartan
  Interventions: Drug: aliskiren; Drug: losartan

INTERVENTIONS:
Drug: aliskiren — Aliskiren will be given in a preliminary dosage of 150 mg per day, after a follow up of two weeks dosage will be increased to 300 mg per day.
Drug: losartan — Losartan will be given in a preliminary dosage of 50 mg per day and after a two weeks follow up dosage will be increased to 100 mg per day

SUMMARY:
Aliskiren is a novel renin inhibitor approved for the treatment of hypertension. The effect of aliskiren on arterial stiffness, inflammation and oxidative stress has not been fully investigated yet.The aim of this study is to investigate the effect of aliskiren on arterial stiffness, platelet function and inflammation compared to losatan in patients with diabetes mellitus.

We hypothesize that aliskiren will have a beneficial effect on arterial stiffness and platelet function in patients with diabetes mellitus.

DETAILED DESCRIPTION:
Background:

Patients with diabetes mellitus (DM) have an increased risk for atherothrombotic events.

Platelets play an important role in cardiovascular disease both in the pathogenesis of atherosclerosis and in the development of acute thrombotic events. Their importance in coronary heart disease is indirectly confirmed by the benefit of antiplatelet agents in these disorders. Platelet adhesion, aggregation and activation are abnormal in patients with DM. Several factors were found to be associated with the abnormalities in platelet signaling in patients with DM, including increased levels of reactive oxygen species, altered calcium mobilization and increased protein tyrosine phosphorylation.

Arterial stiffness, assessed noninvasively by measuring the aortic pulse wave velocity (PWV), is considered a powerful and independent risk factor for early mortality. Increased arterial stiffness may lead to early pulse wave reflection causing an increase in systolic blood pressure and a decrease in diastolic blood pressure. This in turn, increases the myocardial oxygen demand, reduces ejection fraction and increases the left ventricular working load. PWV probably represents an integrated index of vascular structure and function, being influenced by many factors including age, blood pressure, lipid profile and glucose levels. For any level of systolic blood pressure, aortic PWV is found to be increased in diabetic patients compared to nondiabetic patients.

Aliskiren is the first direct renin inhibitor that was introduced for the treatment of hypertension. Aliskiren binds to the active site of renin, inhibiting the activation of the renin- angiotensin- aldosteron (RAAS) system at the rate limiting step. Aliskiren inhibits the conversion of angiotensinogen to angiotensin I (AI). This direct inhibition may be more efficient than the indirect blockade of ACE inhibitors or ARBs.

Except for its BP lowering effect aliskiren was found to increase renal blood flow to a higher degree than that was found for angiotensin converting enzime (ACE) inhibitors or angiotensin receptor blockers (ARBs). Moreover- it blocks the active site of the prorenin/renin ((pro)renin) receptors reducing the local angiotensin II (AII) generation. Renin inhibitors, like the ACE inhibitors or ARBs, increase the concentration of renin which activates the (pro)renin receptors. Renin receptors were found in the kidney, blood vessels and the heart. Binding of renin to these receptors increases its catalytic effect and probably activates a potentially pathogenic, mitogen activated protein kinase pathway. It has a tissue damaging effect by increasing frofibrotic pathways and the expression of molecules such as TGF- beta.

In a recent study aliskiren was found to bind both to renin and prorenin receptors and increase their stability, this rise is probably not causing AII generation although it allows the detection of prorenin as renin. Aliskiren increases the amount of circulating immunoreactive renin but decreases the PRA.

Uresin Y et al compared the efficacy and safety of aliskiren with that of ramipril in patients with diabetes and hypertension. Aliskiren was found to be more effective at lowering systolic blood pressure (SBP) than ramipril, and showed no inferiority in reducing diastolic blood pressure (DBP). When used in combination with ramipril, aliskiren showed a significant additional reduction in both SBP and DBP. In the same study, plasma renin concentration (PRC) was significantly increased with each monotherapy and when combined, PRC increased to a greater level than the sum of the effects of each alone. The reactive rise in PRC was associated with a concomitant rise in plasma renin activity (PRA) in the ramipril group, an effect that was suppressed when combined with aliskiren.

Other recent studies found similar results when comparing efficacy and safety of aliskiren and ramipril or adding it to treatment with valsartan. Safety of aliskiren was also evaluated in elderly patients (above 65) and was found to effectively reduce blood pressure and to be well tolerated in this subgroup of patients.

Inhibition of the RAAS in diabetic patients is known to result in several beneficial effects, independent of their BP lowering effect; Reduction of albumin excretion, prevention of the progression of renal disease and possibly a cardio-protective effect. Valsartan was also found to reduce PWV, and hence arterial stiffness, in diabetic patients independently of its BP lowering effect. Several of these effects had already been evaluated using aliskiren, for example: Nussberger J at al evaluated the effect of aliskiren on atherosclerosis and plaque stabilization in mice, comparing it with atenolol, amlodipine and irbesartan. They found that although they all had a similar blood pressure lowering effect, aliskiren and irbesartan had a beneficial effect on plaque phenotype (including smooth muscle cell content, fibrous cap, lipid core, medial degeneration and macrophage content) whereas amlodipine and atenolol did not. Lu H et al. evaluated the effect of aliskiren on atherosclerosis in LDL receptor deficient mice. They found a significant reduction in atherosclerotic plaque size in the aortic root and arch in the aliskiren treated mice. Aliskiren was found to reduce BP, prevent albuminuria and suppress the renal gene expression of (pro)renin receptors in a model of hypertensive diabetic renal damage in rats. It also exhibited a potential to inhibit prorenin. When using the combination of aliskiren and losartan in patients with DM, aliskiren revealed a reno-protective effect that was independent of its BP lowering effect. The effect of aliskiren on arterial stiffness is yet to be evaluated.

Several studies have evaluated the effect of RAAS system inhibitors on platelet function and hemostasis, for example perindopril was found to have anti-platelet and profibrinolytic effects and telmisartan was found to have anticoagulant effect. Perindopril was also found to reduce platelet aggregation and adrenaline induced platelet aggregation.

The effect of aliskiren on platelet activity is not clear. In an in vitro study biomarkers of platelet activity were not altered by aliskiren (except for a moderate increase of antithrombin-III activity). At higher doses (exceeding its therapeutic range) it had a diverging effect - both platelet activating and antiplatelet effects

Purpose:

The purpose of the study is to evaluate the effect of aliskiren, which inhibits the rate limiting step of the RAAS system, on arterial stiffness, inflammation and platelet function in patients with DM.

Methods:

Study design:

The study will be a prospective, cross over, randomized trial. All patients fulfilling the inclusion and exclusion criteria, after a short screening period, will be treated with aliskiren or losartan. After a washout period of 2 weeks a cross over will be made between the two groups. Aliskiren will be given in a preliminary dosage of 150 mg per day, after a follow up of two weeks dosage will be increased to 300 mg per day. Losartan will be given in a preliminary dosage of 50 mg per day and after a two weeks follow up dosage will be increased to 100 mg per day. Two weeks after initiation of each treatment potassium and creatinin levels will be assessed. The follow up will be conducted in the Research and Development unit in Assaf Harofeh Medical Center at 0, 3 and 6 months and after the wash out period. On each visit patients BP will be assessed by 24 ambulatory BP monitoring. Blood will be drawn (10 cc) for Hemoglobin levels, electrolytes, renal and liver functions, total cholesterol, high density lipoprotein-cholesterol (HDL- cholesterol), triglycerides (TG), oxidized low density lipoprotein (ox-LDL) and hs- CRP. LDL-cholesterol will be calculated. PRA will be measured by radioimmunoassay of generated AI, PRC and plasma aldosterone will be measured by immunochemiluminescence. In addition NO and isoprostane will be measured as an index to oxidative stress. Platelet function and arterial stiffness will be assessed. The patients' medication regimen will not be changed throughout the study period.

Platelet Function Tests Cone-and-Platelet Analyzer 200 µL of citrated blood will be placed in a polystyrene well and subjected to a shear rate of 1300 sec-1 using a rotating conical disk for 2 minutes. The well will be washed and stained by May-Gruenwald stain. Platelet adhesion will be evaluated as the percentage of total area covered with platelets designated as surface coverage (%) and aggregation as the mean size of the surface-bound aggregates designated as average size (µ'm2) by use of an image analysis system (Galai).

Aspirin Response Assay 3.6µl Arachidonic Acid and 0.2 ml blood will be added to a micro tube (2ml), (final Arachidonic Acid concentration 0.275 mM). The tube will be rotated on the tube mixer at 10 rpm for 1 minute. 130 µl will be placed in a well and tested with the cone and platelet analyzer.

Clopidogrel Response Assay 5 µl ADP and 0.2 ml blood will be added into a micro tube (2 ml) (final ADP concentration 1.25 µM). The tube will be rotated on the tube mixer at 10 rpm for 1 minute. 130 µl will be placed in a well and tested with the cone and platelet analyzer. (Varon D et al 1997) Arterial stiffness Assessment of arterial stiffness will be performed by a noninvasive technique using the commercially available SphygmoCor System (AtCor Medical LTD, Australia). All measurements will be performed while the patient is in a recumbent position at a room temperature of 25۫ C, between 06:30 and 08:30 A.M. after an overnight fasti (8-10 hours) and after a short period of rest. Peripheral pressure waveforms will be recorded from the radial artery at the wrist, using applanation tonometry with a high fidelity micromanometer. When sequential waveforms will be recorded, a validated 16-18 generalized transfer function will be applied to generate the corresponding central pressure waveform. The integral system software will be used to calculate an average radial artery waveform and to derive a corresponding central aortic pressure waveform using a previously validated generalized transfer function. From these data the indexes of arterial stiffness will be obtained. The augmentation of central arterial pressure is the difference between the first and second systolic peaks of the central pressure waveforms, and the central augmentation index (AIx) is the augmentation expressed as a percentage of the pulse pressure.

This technology is easy to use, non-invasive, simple, rapid (15 minutes per test) and repeatable.

ELIGIBILITY:
Inclusion Criteria:

* The study will include 40 patients aged 18 years or older with DM, defined as patients with fasting plasma glucose above 126 mg/dL or

  * symptoms of DM with random blood glucose concentration of above 200 mg/dL, or
  * patients treated with oral hypoglycemics or insulin.
* In addition, prior to their enrollment in the study patients' BP will be assessed by 24 hour ambulatory BP monitoring.
* All patients will have to be treated with ACE inhibitors, aspirin and statins for at least one month prior to their enrollment in the study.
* Patients' medication regimen will not be altered during the study period.
* Patients will sign a written informed consent before their inclusion in the study.

Exclusion Criteria:

* Patients will be excluded from the study if their systolic BP is between bellow 110 mmHg or above 150 mmHg mmHg.
* Major exclusion criteria will be:
* acute coronary syndrome in the 6 months previous to the study,
* renal failure with creatinin levels above 1.5 mg/dL,
* hyperkalemia (K > 5 mg/dL),
* hematologic or solid malignancies,
* pregnancy
* a platelet count below 100,000.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
arterial stiffness and platelet function | 6.5 months

SECONDARY OUTCOMES:
oxidative stress parameters (oxidized LDL and Isoprostanes), markers of inflammatory status (highly sensitive CRP test) and 24 hours blood pressure monitoring | 6.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Koren Peleg, MD, Principal Investigator — Department of Internal Medicine A , Research & Development unit Assaf Harofeh Medical Center, Zerifin, affiliated to Sackler School of Medicine, Tel Aviv, Israel